CLINICAL TRIAL: NCT02138227
Title: A Randomized Trial of the Early Referral and Request Approach (ERRA) Intervention to Increase Consent to Organ Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01DK081118 (NIH); 5R01DK081118 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-05-14 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Organ Donation
Keywords: Organ donation request; Effective Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assisted CEaD Condition (Active Comparator): In the assisted condition, participants use the CEaD training materials supplemented with simulators to practice the communication skills.
  Interventions: Behavioral: Assisted CEaD Condition
- Autonomous CEaD Condition (Active Comparator): In the autonomous condition, participants view the CEaD training materials on a DVD along with a self-training guide.
  Interventions: Behavioral: Autonomous CEaD Condition

INTERVENTIONS:
Behavioral: Assisted CEaD Condition — In the assisted condition, participants use the CEaD training materials supplemented with simulators to practice the communication skills. OPO requesters will be assisted by having the CEaD DVD supplemented through working the scenarios with live simulated patients who will be trained to act out the scenarios with the OPO requesters and provide feedback.
  Arms: Assisted CEaD Condition
Behavioral: Autonomous CEaD Condition — In the autonomous condition, participants view the CEaD training materials on a DVD along with a self-training guide.
  Arms: Autonomous CEaD Condition

SUMMARY:
The purpose of this study is to evaluate the efficacy and generalizability of a communication intervention (Communication Effectively about Donation (CEaD)) for Organ Procurement Organization (OPO) staff requesters and to compare two conditions of delivering the CEaD. The experimental design will test: (1) the overall efficacy of the intervention on timely referral and consent for organ donation and (2) whether a completely autonomous condition (no outside training assistance) is clinically equivalent to the assisted condition (training provided by outside consultants) in terms of the final outcome of consent to donation.

DETAILED DESCRIPTION:
For Organ Procurement Organizations (OPO) to be successful, they must be able to obtain consent for organ donation. Despite donor registries, first person consent, and the sharp rise in living donation, transplantation medicine continues to rely on the donation of organs from deceased individuals. Most of these requests are made to the deceased's next of kin. Of all the activities performed by OPOs, obtaining consent to donation is the most important activity as it facilitates all other aspects of the organ procurement and transplantation process. Moreover, communicating with families about the option to donate in a way that provides them with sufficient information to make an informed decision is essential to OPO success in obtaining consent. Our study tested an intervention strategy that addresses this critical aspect of obtaining consent to organ donation.

From 2003 - 2007, we tested the Communicating Effectively about Donation (CEaD) intervention as part of the Early Referral and Request Approach model (ERRA) (HRSA grant # R39 OT01126). The intervention demonstrated significant promise as the analysis of our data indicates an increase in the consent rate of 32.2% and taught OPO staff requesters communication skills that enable them to make effective requests to donor-eligible families. Training involved a series of simulated scenarios, and the intent of the CEaD intervention is to increase the number of organs available for transplantation through improved consent rates by incorporating a systematic approach to training staff for the crucial task of communication about organ donation with family decision-makers.

In our recently completed study (HRSA grant#), we examined the efficacy and generalizability of the CEaD in diverse geographic sites and to compare two conditions of delivering the CEaD. The experimental design tested: (1) the overall efficacy of the CEaD intervention on consent and (2) whether the more cost-saving "autonomous" condition is clinically equivalent to the "assisted" condition in terms of the final outcome of consent to donation. The major outcome measures were: 1) success in achieving relational communication with donor families and, 2) consent to donation.

The major goals of this study were to provide OPOs with the tools to assess and train OPO staff on a sustained basis. Specifically, we:

1. Packaged the CEaD as a self-teach tool so that OPOs can provide basic and continuous training for OPO staff requesters in the use of effective communication techniques when making requests to donor-eligible families.
2. Tested the effectiveness of the CEaD training program to increase consent rates, regardless of implementation condition, in a sample of OPOs. Our sub-hypotheses included the following:

   H2a: When compared to the 12 month pre-intervention control period, the post-intervention period (after implementation of the CEaD) would be associated with a greater percentage of requests that use the preferred communication techniques with donor-eligible families.

   H2b: When compared to the control period, the overall consent rate during the post-intervention period will be significantly greater than the consent rate during the control period.
3. Tested whether OPOs are able to implement the CEaD assessment and training intervention using two methods for implementation. The two implementation methods tested were: 1) a completely autonomous method in which the OPO does not employ any outside assistance to implement the module, and 2) an assisted method whereby trained outside consultants play a role in helping the OPO implement the CEaD. OPOs will be randomized to one of these two conditions: 1) autonomous CEaD; and 2) assisted CEaD.

H3a: The autonomous CEaD implementation groups will not be as effective as the assisted CEaD implementation groups as measured by preferred communication techniques with donor-eligible families.

H3b: The autonomous CEaD implementation group will not be as effective as the assisted CEaD implementation groups when controlling for the method of delivery for CEaD as measured by consent rates.

The study 'subjects' included the 9 OPOs and their staff (n=273) who make requests to families of deceased donor-eligible patients (termed 'OPO Requesters'). All OPO staff who request organs from families were invited to participate in the study. We obtain written informed consent from each participating requester before we administered surveys. Each survey instrument reminded OPO staff that they are free to withdraw from the study at any time and that the information provided by them was kept strictly confidential. Using a random number generator, requesters were randomized on the OPO level to account for the differences in OPO size, scope, and organizational structure. A total of 218 requesters were randomized to the autonomous condition, and 55 were randomized to the assisted condition.

Intervention The intervention tested two methods of using the Communicating Effectively about Donation (CEaD) intervention. The CEaD taught OPO staff requesters communication skills using a series of simulated scenarios and was designed to allow requesters to make effective requests to donor-eligible families. The training materials were made available on a secure website (www.ceadtraining.org; user name: test; password: test). We compared two methods of training: 1) using the training materials supplemented with simulators to practice the communication skills (assisted) or, 2) viewing the training materials along with a workbook (autonomous). The purpose of this design was to ascertain whether OPOs are capable of successfully employing the CEaD training program on their own, without incurring the added cost of hiring outside consultants.

Description of the Communicating Effectively about Donation (CEaD) Training Program The CEaD intervention was not just a generic communications intervention, but one specifically and uniquely tailored to the problem of making requests for organ donation to families of deceased patients. The intervention was also designed to provide OPO requesters a basic framework for the request conversation. The CEaD trains requesters to make effective requests to donor-eligible families by allowing requesters to learn and practice relational communication skills using a series of scenarios. These scenarios, created in consultation with our partner OPO, involved the use of simulated patients (SPs), who played the role of bereaved family members faced with the opportunity to donate a loved one's organs. Based on our previous study, we developed four training scenarios, the first an uncomplicated scenario, the second an African-American family, the third a pediatric patient whose parents are divorced and at odds, and the fourth a donation after cardiac death (DCD) case. Each scenario allows the requester to use basic requester skills including framing donation positively, using statistics to explain donation benefits, engaging the family in a discussion of their values, probing and responding to family fears or misinformation about donation, and attending to family's emotional needs. The scenarios also allowed requesters to work through increasingly more challenging donation situations and to encounter specific issues such as the dysfunctional family, minority families, and families whose opinions about whether or not to donate are divided.

The scenarios focused on training requesters to use the following communication skills:

(1) assessing families' and patients' beliefs and values regarding organ donation; (2) assessing families' readiness to hear about organ donation; and, (3) using communication skills, such as listening, responding empathetically, and dealing with ambivalence, when dealing with grieving families.

ELIGIBILITY:
Inclusion Criteria:

* OPO requester staff employed at a participating OPO
* Family decision makers (FDM) approached by a participating OPO requester about the option of donating the organs of their loved one
* 16 years of age or older (16 and 17 year old FDM will require consent of custodial adult)

Exclusion Criteria:

* OPO requester staff not employed at a participating OPO
* FDM not approached by a participating OPO requester
* FDM younger than 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Siminoff, PhD, Principal Investigator — Temple University; Heather M Traino, PhD, Principal Investigator — Virginia Commonwealth University
Locations (9):
- United States (9):
  - Alabama Organ Center, Birmingham, Alabama
  - Donor Network of Arizona, Phoenix, Arizona
  - TransLife of Orlando, Winter Park, Florida
  - New England Organ Bank, Waltham, Massachusetts
  - Mid-America Transplant Services, Springfield, Missouri
  - New York Organ Donor Network, New York, New York
  - LifeBanc, Cleveland, Ohio
  - LifeGift Organ Donation Center, Houston, Texas
  - LifeNet, Richmond, Virginia

REFERENCES:
- [Result] Traino HM, Siminoff LA. Attitudes and acceptance of First Person Authorization: a national comparison of donor and nondonor families. J Trauma Acute Care Surg. 2013 Jan;74(1):294-300. doi: 10.1097/TA.0b013e318270dafc. PMID 23147186
- [Derived] Siminoff LA, Alolod GP, Gardiner HM, Hasz RD, Mulvania PA, Wilson-Genderson M. A Comparison of the Content and Quality of Organ Donation Discussions with African American Families Who Authorize and Refuse Donation. J Racial Ethn Health Disparities. 2021 Apr;8(2):485-493. doi: 10.1007/s40615-020-00806-7. Epub 2020 Jun 30. PMID 32607720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: While 273 participants registered, data were used from only 134 subjects, who had encounters pre- and post-intervention.
Period: Overall Study
Arm/Group | Assisted CEaD Condition | Autonomous CEaD Condition
Started | 55 | 218
Completed | 55 | 218
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assisted CEaD Condition | Autonomous CEaD Condition | Total
Number analyzed (Participants) | 55 | 218 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.72 (9.96) | 44.42 (9.46) | 44.88 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 161 | 197
  Male | 19 | 57 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Authorization Rates for Solid Organ Donation From Families of Donor-eligible Patients
Description: OPO requesters completed a brief, web-based survey after every family approach, regardless of whether the family ultimately consented to donation. Rates of baseline and post-intervention consent to donation were compared. Due to the repeated measures design of the study and the high turnover rate among requesters, the number of participants in the post-intervention arms will not sum to those in the corresponding pre-intervention tenure level.
Time Frame: Baseline and continuously for 3 years post intervention
Measure: Number; unit: Percentage of successful requests
Units Other Than Participants: Total organ donation approach encounters
Groups:
- Pre-Intervention Authorization Rate (All Novice): This is the authorization rate (successful authorization requests/total authorization requests) of participants in aggregate before the intervention. Novice participants are defined has having less than 12 months of experience.
- Post-Intervention Authorization Rate (Novice Autonomous Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the autonomous arm after the intervention. Novice participants are defined has having less than 12 months of experience.
- Post-Authorization Rate (Novice Assisted Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the assisted arm after the intervention. Novice participants are defined has having less than 12 months of experience.
- Pre-Intervention Authorization Rate (All Mid-Level): This is the authorization rate (successful authorization requests/total authorization requests) of participants in aggregate before the intervention. Mid-level participants are defined has having 13 to 36 months of experience.
- Post-Intervention Authorization Rate(Mid-Level Autonomous Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the autonomous arm after the intervention. Mid-level participants are defined has having 13 to 36 months of experience.
- Post-Authorization Rate (Mid-Level Assisted Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the assisted arm after the intervention. Mid-level participants are defined has having 13 to 36 months of experience.
- Pre-Intervention Authorization Rate (All Senior): This is the authorization rate (successful authorization requests/total authorization requests) of participants in aggregate before the intervention. Senior participants are defined has having more than 36 months of experience.
- Post-Intervention Authorization Rate (Senior Autonomous Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the autonomous arm after the intervention. Senior participants are defined has having more than 36 months of experience.
- Post-Authorization Rate (Senior Assisted Arm): This is the authorization rate (successful authorization requests/total authorization requests) of participants in the assisted arm after the intervention. Senior participants are defined has having more than 36 months of experience.
Arm/Group | Pre-Intervention Authorization Rate (All Novice) | Post-Intervention Authorization Rate (Novice Autonomous Arm) | Post-Authorization Rate (Novice Assisted Arm) | Pre-Intervention Authorization Rate (All Mid-Level) | Post-Intervention Authorization Rate(Mid-Level Autonomous Arm) | Post-Authorization Rate (Mid-Level Assisted Arm) | Pre-Intervention Authorization Rate (All Senior) | Post-Intervention Authorization Rate (Senior Autonomous Arm) | Post-Authorization Rate (Senior Assisted Arm)
Number analyzed (Participants) | 31 | 30 | 10 | 27 | 15 | 6 | 45 | 22 | 12
Number analyzed (Total organ donation approach encounters) | 144 | 192 | 137 | 158 | 101 | 51 | 266 | 170 | 129
Percentage of successful requests | 78 | 80 | 89 | 81 | 76 | 88 | 89 | 92 | 83

2. Secondary Outcome: Change in Requesters' Aggregated Relational Communication Skills
Description: Using a family interview, we will examine the family's experience with the donation process, specifically focusing on family self-report of comfort, satisfaction with the communication and decision-making process, content of the conversation, and measurement of the relational aspects of the communication. The instrument is based on a well-developed interview that was used in a seminal study of family experience and decision-making for organ donation in acute care hospital settings. Due to the repeated measures design of the study and the high turnover rate among requesters, the number of participants in the post-intervention arms will not sum to those in the corresponding pre-intervention tenure level. The aggregate scores of fourteen (14) 7-point scale items with an aggregate range of 14 to 98. Higher values represent a better outcome.
Time Frame: Baseline and continuously for 3 years post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Total organ donation approach encounters
Groups:
- Novice Pre-Intervention Aggregate Relational Communication: Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of novice requesters pre-intervention. Novice participants are defined has having less than 12 months of experience.
- Novice Post-Intervention Relational Communication (Autonomous): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of novice requesters from the autonomous arm. Novice participants are defined has having less than 12 months of experience.
- Novice Post-Intervention Relational Communication (Assisted): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of novice requesters in the assisted arm. Novice participants are defined has having less than 12 months of experience.
- Mid-Level Pre-Intervention Aggregate Relational Communication: Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of mid-level requesters pre-intervention. Mid-level participants are defined has having 13 to 36 months of experience.
- Mid-Level Post Intervention Relational Com (Autonomous): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of mid-level autonomous post-intervention autonomous arm. Mid-level participants are defined has having 13 to 36 months of experience.
- Mid-Level Post-Intervention Relational Com (Assisted): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of mid-level requesters in the autonomous post-intervention arm. Mid-level participants are defined has having 13 to 36 months of experience.
- Senior Pre-Intervention Aggregate Relational Communication: Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of senior requesters pre-intervention. Senior participants are defined has having more than 36 months of experience.
- Senior Post-Intervention Relational Communication (Autonomous): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of senior requesters in the autonomous post-intervention arm. Senior participants are defined has having more than 36 months of experience.
- Senior Post-Intervention Relational Communication (Assisted): Mean of items measuring emotion, tone, and levels of sincerity, honesty, willingness to listen, and cooperation of senior requesters in the assisted post-intervention arm. Senior participants are defined has having more than 36 months of experience.
Arm/Group | Novice Pre-Intervention Aggregate Relational Communication | Novice Post-Intervention Relational Communication (Autonomous) | Novice Post-Intervention Relational Communication (Assisted) | Mid-Level Pre-Intervention Aggregate Relational Communication | Mid-Level Post Intervention Relational Com (Autonomous) | Mid-Level Post-Intervention Relational Com (Assisted) | Senior Pre-Intervention Aggregate Relational Communication | Senior Post-Intervention Relational Communication (Autonomous) | Senior Post-Intervention Relational Communication (Assisted)
Number analyzed (Participants) | 31 | 30 | 10 | 27 | 15 | 6 | 45 | 22 | 12
Number analyzed (Total organ donation approach encounters) | 144 | 192 | 137 | 158 | 101 | 51 | 266 | 170 | 129
units on a scale | 75.22 (7.6) | 77.7 (7.8) | 78.0 (7.4) | 75.60 (9.0) | 75.0 (9.0) | 77.0 (7.3) | 76.10 (7.7) | 76.13 (7.7) | 78.2 (7.4)
Statistical Analysis 1: Comparison: Novice Pre-Intervention Aggregate Relational Communication; Test type: Superiority or Other; p < 0.01, ANOVA

3. Secondary Outcome: Change in Request Staff's Comfort Answering Donation-related Questions During the Approach to Family Decision Makers
Description: Requester staff self-report assessment utilizing a seven-point scale to rate his/her own comfort and satisfaction with the overall request process following each family contact. Due to the repeated measures design of the study and the high turnover rate among requesters, the number of participants in the post-intervention arms will not sum to those in the corresponding pre-intervention tenure level. The assessment was performed using a Likert scale ratin with a range of 1 to 7, with higher values representing better outcomes.
Time Frame: Baseline and continuously for 3 years post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Organ Donation Encounters
Groups:
- Novice Pre-Intevention Aggregate Requester Comfort: Mean level of comfort with novice staff self-reported pre-intervention. Novice participants are defined has having less than 12 months of experience.
- Novice Post-Intervention Requester Comfort (Autonomous): Mean level of comfort novice staff self-reported post- intervention in the autonomous arm. Novice participants are defined has having less than 12 months of experience.
- Novice Post-Intervention Requester Comfort (Assisted): Mean level of comfort novice staff self-reported post-intervention in the assisted arm. Novice participants are defined has having less than 12 months of experience.
- Mid-Level Pre-Intervention Aggregate Requester Comfort: Mean level of comfort mid-level staff self-reported pre-intervention. Mid-level participants are defined has having more 13 to 36 months of experience.
- Mid-Level Post-Intervention Requester Comfort (Autonomous): Mean level of comfort mid-level staff self-reported post-intervention in the autonomous arm. Mid-level participants are defined has having more 13 to 36 months of experience.
- Mid-Level Post-Intervention Requester Comfort (Assisted): Mean level of comfort mid-level staff self-reported post-intervention in the assisted arm. Mid-level participants are defined has having more 13 to 36 months of experience.
- Senior Pre-Intevention Aggregate Requester Comfort: Mean level of comfort senior staff self-reported pre-intervention. Senior participants are defined has having more than 36 months of experience.
- Senior Post-Intervention Requester Comfort (Autonomous): Mean level of comfort senior staff self-reported post-intervention in the autonomous arm. Senior participants are defined has having more than 36 months of experience.
- Senior Post-Intervention Requester Comfort (Assisted): Mean level of comfort senior staff self-reported post-intervention in the assisted arm. Senior participants are defined has having more than 36 months of experience.
Arm/Group | Novice Pre-Intevention Aggregate Requester Comfort | Novice Post-Intervention Requester Comfort (Autonomous) | Novice Post-Intervention Requester Comfort (Assisted) | Mid-Level Pre-Intervention Aggregate Requester Comfort | Mid-Level Post-Intervention Requester Comfort (Autonomous) | Mid-Level Post-Intervention Requester Comfort (Assisted) | Senior Pre-Intevention Aggregate Requester Comfort | Senior Post-Intervention Requester Comfort (Autonomous) | Senior Post-Intervention Requester Comfort (Assisted)
Number analyzed (Participants) | 31 | 30 | 10 | 27 | 15 | 6 | 45 | 22 | 12
Number analyzed (Organ Donation Encounters) | 144 | 192 | 137 | 158 | 101 | 51 | 266 | 170 | 129
units on a scale | 4.91 (0.33) | 6.88 (0.41) | 6.89 (0.66) | 6.79 (0.66) | 6.99 (0.14) | 6.91 (0.30) | 6.80 (0.74) | 6.98 (0.21) | 6.98 (0.19)
Statistical Analysis 1: Comparison: Novice Pre-Intevention Aggregate Requester Comfort; Test type: Superiority or Other; p < 0.01, ANOVA; F (2, 1574)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Assisted CEaD Condition | Autonomous CEaD Condition
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/218
Other Adverse Events (participants affected / at risk) | 0/55 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes